CLINICAL TRIAL: NCT03336762
Title: Injured Spinal Cord Pressure Evaluation Study - Transverse Myelitis
Acronym: ISCoPE-TM
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: Wings for Life (Other); Neurosciences Research Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16.0089
Record Dates: First submitted 2017-11-01; First posted 2017-11-08 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Transverse Myelitis
MeSH Terms: conditions — Myelitis, Transverse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Intra spinal pressure monitoring — Sub dural pressure monitoring using a FDA approved intracranial pressure monitor
Diagnostic Test: Intra spinal microdialysis monitoring — Sub arachnoid microdialysis monitoring using a FDA approved hepatic microdialysis catheter

SUMMARY:
ISCoPE-TM will use intra spinal monitoring techniques to assess cord perfusion and metabolism in patients with severe spinal cord damage from transverse myelitis

DETAILED DESCRIPTION:
Transverse myelitis (TM) is a rare inflammatory condition of the spinal cord. It is characterised by rapid onset of motor, sensory or autonomic dysfunction causing neurological deficit. It has a diverse range of causes; most commonly it is associated with multiple sclerosis and neuromyelitis optica also known as Devic's disease or Devic's syndrome, is a heterogeneous condition consisting of the simultaneous inflammation and demyelination of the optic nerve (optic neuritis) and the spinal cord (myelitis). It affects approximately 1900 adults and children in the UK annually, with 350 cases per year of unknown cause.

Outcome in TM is variable; e.g. neuromyelitis optica mortality can be 30% . There is a relationship between the severity of neurological symptoms at presentation and the eventual outcome. When a patient is ASIA (American spinal injuries association) A or tetraplegic at presentation, they are less likely to recover than when ASIA B/C or paraplegic. Approximately 30% of patients will be ASIA A-C after a TM episode.

There are several pathological mechanisms which could increase the risk of decreased blood supply and further neurological deficit in TM. The ISCoPE study has shown that in traumatic spinal cord injury when swelling causes mechanical compression of the cord against the dura there is increased intra spinal pressure (ISP).

The Investigators propose to monitor the ISP and spinal cord metabolites in 10 TM patients with MRI evidence of a swollen enlarged spinal cord. There has never been a study looking at ISP in TM patients before. The optimum blood pressure in patients with TM is not known.

The investigators aim to observe a previously unrecognised pathological mechanism of injury in TM. In the future this could lead on to novel treatments to improve drug delivery and neurological outcome in a condition otherwise associated with a poor outcome.

ELIGIBILITY:
Inclusion Criteria:

* Transverse myelitis (as defined by TM working group 2002)
* MRI evidence of swollen enlarged spinal cord. Defined as a larger cord diameter compared to the adjacent normal signal intensity spinal cord, with loss of cerebrospinal fluid space between cord and dura mater.
* Age 18 - 70
* Severe spinal cord injury (ASIA A - B)
* Monitoring to start within 72 h of MRI
* Capacity for informed consent

Exclusion Criteria:

* Major co-morbidities likely to influence outcome
* High anaesthetic risk precluding surgery
* Multiple separate lesions on MRI spine
* Lacking capacity or Unable to consent
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with formal diagnosis of transverse myelitis
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events as assessed by CTCAE v4.0 | Through study completion, up to 1 year.
  To assess whether intraspinal pressure and metabolism monitoring in Transverse Myelitis patients is feasible and safe

SECONDARY OUTCOMES:
Intra spinal pressure in mmHg | Up to 7 days
  To determine whether the swollen, enlarged spinal cord in patients with transverse myelitis causes raised intra spinal pressure, low spinal cord perfusion pressure
Injury site metabolism measured using surface microdialysis. | Up to 7 days
  To determine whether the swollen, enlarged spinal cord in patients with transverse myelitis causes deranged spinal cord metabolites (glucose, lactate, pyruvate, glycerol, glutamate)

CONTACTS AND LOCATIONS:
Overall Officials: Marios Papadopoulos, MD, Principal Investigator — St George's, University of London
Locations (1):
- St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No